CLINICAL TRIAL: NCT04646356
Title: Tacrolimus Trial for Hereditary Hemorrhagic Telangiectasia (HHT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170518448
Record Dates: First submitted 2020-10-20; First posted 2020-11-27 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Hereditary Hemorrhagic Telangiectasia; Epistaxis Nosebleed
Keywords: Hereditary Hemorrhagic Telangiectasia; HHT; Tacrolimus
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tacrolimus immediate-release capsules (Experimental): subjects will be treated with a 6 months course of oral low-dose tacrolimus capsules to be taken twice daily starting dose of 0.025 mg/kg/day, adjusted to maintain drug blood levels of 2-5ng/ml
  Interventions: Drug: Tacrolimus capsule (low-dose)

INTERVENTIONS:
Drug: Tacrolimus capsule (low-dose) — low-dose Tacrolimus will be given for 6 months followed by a washout period for 6 months

SUMMARY:
This study will investigate the effectiveness of oral low-dose tacrolimus for the treatment of recurrent nasal hemorrhage in HHT subjects. The primary outcome for the trials will be the reduction of epistaxis severity (minutes of bleeding per week). The biological outcomes of interest are the regression of vascular malformations as well as tissue and circulation biomarkers of the relevant mechanistic pathways. In this Phase II open label trial, we estimate a sample size of 30 subjects with HHT, with moderate-severe recurrent epistaxis will be required. Subject will be treated with a 6-month course of tacrolimus twice daily.

DETAILED DESCRIPTION:
The aim is to study is to evaluate low-dose tacrolimus as a treatment for HHT. Rare disease presents a number of challenges in clinical trial design, including recruitment challenges, related power limitations and less knowledge about outcomes measurement. Considering these limitations, as well as the large variability in epistaxis measures across HHT patients, a trial design, with each subject receiving the study drug for six months and for one year an epistaxis daily dairy documentation, providing valuable information about seasonal variation.in epistaxis.

This study will investigate tacrolimus, given its demonstrated anti-angiogenic and anti-inflammatory properties, as well as compelling effects in arteriovenous malformation (AVM) models. Specifically, tacrolimus has been shown to oppose the gene expression upregulation of the identified pro-angiogenic markers, thus resulting in anti-angiogenic effects. There are two mechanisms to this. Firstly, recent evidence has shown tacrolimus to be a potent ALK1 signaling mimetic at the transcriptional level. This is particularly significant given that the ALK1 pathway signaling is lost in HHT via the hallmark ACVRL1 and ENG genes. Independent of its effect on the ALK1 pathway, tacrolimus has been shown to be a potent inhibitor of VGEF signaling.

As mentioned previously, the BMP9-ALK1-endoglin-Smad1/5/9 pathway in HHT, is a novel avenue of interest for treating hemorrhage in HHT and also regressing vascular malformations. Given the upstream inactivation of the ALK1 pathway, therapeutic potential via this pathway is dependent on Smad1/5/8 activation and signaling irrespective of the functional status of the corresponding ALK1 receptors. To this end, tacrolimus has been shown to activate Smad1/5/8 signaling in HHT patient-derived cells, thus confirming its therapeutic potential in HHT.

Tacrolimus also has anti-inflammatory effects, via inhibition of pro-inflammatory cytokines, specifically IL2, which is associated with cytotoxic T cell proliferation and activation. Finally, recent evidence also demonstrated a reduction of vascular pathology in mouse models via tacrolimus administration. Tacrolimus also has the advantages of a proven safety track record for long-term use, given its long history in transplant medicine, and can be orally administered, making it more acceptable to patients. In addition to promising effects in laboratory-based studies, Canadian case study reported the regression of angiodysplasia and reduction of mucosal hemorrhage in a probable HHT patient who underwent liver transplantation following high-output cardiac failure and hepatic AVM development. A recent case report of treatment with oral low-dose -dose tacrolimus in an individual with HHT, found that tacrolimus dramatically improved epistaxis. Based on the evidence to date, the investigators hypothesize that oral low-dose tacrolimus will reduce nasal hemorrhage in HHT subjects, through anti-angiogenic and/or anti-inflammatory mechanisms, both of which have been implicated in HHT.

This clinical trial of oral low-dose tacrolimus (0.025mg/kg/day and adjusted to maintain blood levels of 2-5ng/ml 6-month course) in HHT subjects with moderate-severe recurrent nasal hemorrhage. Drug dosing and safety monitoring will be tailored specifically to the agent studied. The primary outcome will be reduction of bleeding minutes per week. In addition, vascular malformation tissue (cutaneous) will be obtained pre and post-investigational product from some subject, and stained for inflammatory, angiogenic and BMP9-ALK1-endoglin- SMAD1/5/9 pathway markers. In addition, pre-excision, vascular malformations will be imaged with speckle variance optical coherence tomography (SVOCT), in vivo non-invasive micro-angiography, to measure lesion structure, vessel volume and vessel density, as previously described. Tissue and imaging may provide important insights into physiological mechanisms that explain clinical changes. If the drugs studied are effective at reducing nasal hemorrhage, this will have important clinical implications for HHT patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Clinical HHT diagnosis or personal genetic diagnosis of HHT
3. Epistaxis at least 15 min per week (mean for past month)
4. At least one telangiectasia (skin or mucosal) available for micro-imaging.
5. Ability to give written informed consent, including compliance with the requirements of the study.

Exclusion Criteria:

1. Allergy/intolerance to the study drug or related agents
2. Unstable medical illness
3. Acute infection
4. Creatinine > ULN (upper limit of normal)
5. Liver transaminases (AST or ALT) >= 2x ULN
6. Women participant who are pregnant or breastfeeding or plan to become pregnant during the duration of the study
7. Women of childbearing potential not on effective contraception. Male participants of reproductive potential whose female partners are of childbearing potential and are not planning to use highly effective contraceptive method
8. BHCG level <6 IUL (re-test if 6-24 IU/L)
9. Specific contra-indications for study drug (detailed in the product monograph)
10. Abnormal ECG where the QTc >480msec

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
The change in epistaxis (nose bleeding) severity using low-dose Tacrolimus | 96 weeks
  Participants will be asked to maintain a daily diary for the duration of the study (96 weeks). Participants will record all epistaxis events daily, noting the duration in minutes and whether or not there was gushing during each nosebleed. The change in epistaxis severity will be measured from a sum of duration of all bleeding events each week, as measured from the participant daily diary.

SECONDARY OUTCOMES:
Change in Epistaxis Severity Score (ESS) | Baseline, Weeks; 12,18,24,30,36,42,48,60,66,72,78,84,96
  The epistaxis severity score is a six item questionnaire used to calculate a severity of HHT related nose bleeding. Each question is pertaining to the subject's typical symptoms within the last 3 months period. The first three questions are related to frequency, duration and intensity. The forth question whether or not medical attention was sought for nose bleeding. The remaining two questions are related to the presence of anemia and the need for blood transfusion due to nose bleeding. The resulting epistaxis severity score vary between; none 0-1, mild bleeding >1-4, moderate bleeding >4-7 and >7-10 for severe bleeding. The ESS questionnaire will be administered to participants at every clinic visit throughout the 96 weeks of the study.
Change in Chronic Bleeding | Baseline, Weeks; 12,18,24,30,36,42,48,60,66,72,78,84,96
  Blood samples will be taken to measure change in chronic bleeding as a safety measure. Samples will be taken prior to investigational product for a baseline value. This will be followed by measurements every six weeks during the periods of investigational product for comparative analysis
Micro-Imaging to measure regression of Vascular Malformations | week 12, week 36, week 60, week 84
  Telangiectases will be micro-imaged using an established medical imaging technique speckle variance optical coherence tomography (SVOCT). The micro-imaging will be used for vasculature measurements and structural images of the telangiectases.
The use of Telangiectasia tissue sample to look at the mechanisms of action of Tacrolimus | week 36, week 84
  A punch biopsy of one cutaneous telangiectasia will be performed at two time points during the study. The biopsy tissue sample will be taken at the end of each 6 month active comparator treatment. The tissue will be analyze and stained for inflammatory, angiogenesis and BMP9-ALK1-endoglin-Smad1/5/9 pathway markers (VEGF, MMP-9, COX-2, Endoglin, ALK1 ) before and after treatment with Tacrolimus
Change in Biomarkers | Weeks: 12, 24, 36, 48, 60, 72, 84, 96
  In order to understand the mechanisms of Tacrolimus effects on vascular malformations and hemorrhage in HHT a serum/plasma sample will be collected before and after treatment with Tacrolimus to measure inflammatory, angiogenesis and BMP9-ALK1-endoglin-Smad1/5/9 pathway markers (VEGF, MMP-9, Thrombospondin-2, ESR, CRP, endothelin)

CONTACTS AND LOCATIONS:
Overall Officials: Marie E Faughnan, MD,MSc,FRCPC, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No